CLINICAL TRIAL: NCT06949228
Title: Adjunctive Intra-arterial Tenecteplase Following Mechanical Thrombectomy (ALLY) II Trial
Acronym: ALLY II TNK
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLY II
Record Dates: First submitted 2025-04-17; First posted 2025-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Acute Disease
Keywords: Stroke; TNK; Thrombolytic
MeSH Terms: conditions — Ischemic Stroke; Acute Disease; Stroke | interventions — Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Randomized to Intra Arterial (IA) Tenecteplase (TNK) (Experimental): Patients will receive IA- TNK
  Interventions: Drug: tenecteplase
- Randomized to best medical practice (No Intervention): Patients will receive best medical practice treatment

INTERVENTIONS:
Drug: tenecteplase — Patients treated with standard of care mechanical thrombectomy (MT) that achieved mTICI 2b or higher revascularization. Patients will be randomized into one of two arms: IA TNK or control.
  Arms: Randomized to Intra Arterial (IA) Tenecteplase (TNK)

SUMMARY:
The study objective is to evaluate the safety and efficacy of Intra arterial (IA) Tenecteplase (TNK) as an adjunctive therapy in acute ischemic stroke (AIS) patients with large vessel occlusions (LVO) in the anterior circulation of Internal Carotid Artery (ICA), Middle Cerebral Arteries (M1 and M2) who achieve a reperfusion grade of Modified Treatment in Cerebral Ischemia Scale (mTICI) 2b or higher post-mechanical thrombectomy using Food and Drug Administration (FDA) approved devices.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Anterior circulation ischemic stroke symptoms with confirmed occlusion (ICA, M1, or M2) on angiogram and mechanical thrombectomy initiated within 24 hours since last known well
3. Alberta Stroke Program Early CT Score (ASPECTS) Score ≥6 on baseline Non-contrast Head CT (NCCT)
4. Post-mechanical thrombectomy with ≤5 device passes and mTICI grade 2b or higher.
5. Ability to obtain signed informed consent prior to randomization from LAR or Subject

Exclusion Criteria:

1. Premorbid modified Rankin scale (mRS) score >1
2. Imaging evidence of hemorrhage or mass effect at baseline
3. Platelet count <100,000
4. Active hemorrhagic diathesis, or known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
5. Active anticoagulation treatment with novel oral anticoagulant (NOACs) taken within the last 48 hours, or INR >1.7
6. Patients requiring active treatment with dual antiplatelet agents (e.g. proximal cervical carotid artery stenting)
7. Pregnant or lactating
8. Previous known allergy to TNK
9. Major surgery in past 30 days
10. Patient is on or requires dialysis
11. History of intracranial hemorrhage or serious head trauma at any time
12. Any condition in the opinion of the enrolling physician that would preclude the patient from participating
13. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional evaluation
14. Severe, uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) that is refractory to treatment
15. History of acute ischemic stroke in the last 60 days and/or has received previous treatment with a thrombolytic within the last 90 days
16. Presumed septic embolus; suspicion of bacterial endocarditis
17. Suspicion of aortic dissection
18. Intracranial neoplasm
19. Any terminal medical condition with life expectancy less than 6 months
20. Concurrent enrollment in another trial that could confound the results of this study
21. Patient is unlikely to return for 90-day follow-up.
22. Intravenous tissue plasminogen activator (tPA) administered concurrently with Intra-arterial TNK

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint- Modified Rankin Scale (mRS) | 90 days (+/- 30 days) post treatment.
  Proportion of patients with Modified Rankin Scale (mRS) 0-1 at 90-days. The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Primary Safety Endpoint- Incidence of Intracranial hemorrhage and Neurologic Worsening | 24 hours (+/-12 hours) post treatment.
  Incidence of any intracranial hemorrhage and neurologic worsening of at least 4 points on the National Institute of Health Stroke Scale (NIHSS) associated with a Parenchymal hematoma, Type 2 (PH2) brain hemorrhage, according to the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) criteria, within 24 (±12) hours from randomization.

SECONDARY OUTCOMES:
Ordinal Modified Rankin Scale (mRS) | 90 days (+/-30 days) post treatment.
  Ordinal mRS at 90 day. The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Functional Independence | 90 days (+/- 30 days) post treatment.
  Proportion of patients with functional independence, defined as a mRS of 0-2 at 90 days.
Final Revascularization Grade | Immediate post treatment.
  Final revascularization grade at end of IA treatment among those with less than mTICI 3 prior to IA-TNK administration.
Mortality rate at 90 days | Mortality rate at 90-days (+/- 30 days) post treatment.
  Mortality rate at 90-days
Mortality Rate at discharge | Day 6 (+/-1 day) or Discharge post treatment.
  Mortality rate at discharge.
Infarct Volume Post Procedure | 24 hours (+/- 12 hours) post treatment.
  Infarct volume on post-procedure follow-up scans performed at 24 ± 12 hours following mechanical thrombectomy.
Asymptomatic Intracranial hemorrhage | 24 hours (+/- 12 hours) post treatment.
  Incidence of any asymptomatic intracranial hemorrhage
Mean Number of Boluses | Immediate post procedure.
  Mean number of boluses to achieve improvement in reperfusion to mTICI 2c and mTICI 3 among those without mTICI3 prior to IA-TNK administration.

CONTACTS AND LOCATIONS:
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zaidi SF, Castonguay AC, Zaidat OO, Jadhav AP, Sheth SA, Haussen DC, Nguyen TN, Burgess RE, Alhajala HS, Gharaibeh K, Salahuddin H, Rao R, Oliver MJ, Jumaa MA. Safety of Adjunctive Intraarterial Tenecteplase Following Mechanical Thrombectomy: The ALLY Pilot Trial. Stroke. 2025 Feb;56(2):355-361. doi: 10.1161/STROKEAHA.124.048846. Epub 2025 Jan 8. PMID 39772606